CLINICAL TRIAL: NCT01861574
Title: Transcranial Magnetic Stimulation (TMS) Effects on Pain Perception
Brief Title: Transcranial Magnetic Stimulation Effects on Pain Perception
Acronym: TMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: HR 15330
Record Dates: First submitted 2012-04-26; First posted 2013-05-23 (Estimated); Results first posted 2018-08-23 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-08

CONDITIONS: Gastric Bypass Surgery Pain Management

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Both Real TMS (Experimental): Participants in the Both Real TMS group receive 20 minutes of Real TMS 45 minutes after gastric-bypass surgery and then another 20 minutes of Real TMS 4 hours after surgery.
  Interventions: Device: Real TMS 45 min; Device: Real TMS 4 Hours
- Sham then Real TMS (Sham Comparator): Participants in the Sham then Real TMS group, receive Sham TMS 45 minutes after gastric-bypass surgery and 20 minutes of Real TMS 4 hours after surgery.
  Interventions: Device: Sham TMS 45 min; Device: Real TMS 4 Hours
- Real then Sham TMS (Sham Comparator): Participants in the Real then Sham TMS group receive 20 minutes of Real TMS 45 minutes after gastric-bypass surgery and then 20 minutes of Sham TMS 4 hours after surgery.
  Interventions: Device: Real TMS 45 min; Device: Sham TMS 4 Hours
- Both Sham TMS (Sham Comparator): Participants in the Both Sham TMS group, receive Sham TMS 45 minutes after gastric-bypass surgery and then another 20 minutes of Sham TMS 4 hours after surgery
  Interventions: Device: Sham TMS 45 min; Device: Sham TMS 4 Hours

INTERVENTIONS:
Device: Real TMS 45 min — Real TMS 45 minutes after surgery, first determined resting motor threshold (rMT) by starting with 40% of the machine output and 0.5 Hz stimulus frequency. The coil was positioned over the motor cortex and then adjusted until each pulse results in movement of the right thumb. The machine output was then adjusted to the lowest intensity that reliably produces thumb movement. Parameter estimation by sequential testing was used to determine the amount of machine energy necessary to visibly move the thumb 50% of the time. rMT was assessed before each rTMS treatment. The left prefrontal cortex was the cortical target for rTMS treatment. The EEG-10-20 system was used to locate the prefrontal cortex (F3).
  Other Names: NeoPulse Neotonus Model 3600
  Arms: Both Real TMS; Real then Sham TMS
Device: Sham TMS 45 min — Sham TMS 45 minutes after surgery used specifically designed rTMS coil that produces auditory signals identical to real (active) TMS coils but is shielded so that actual stimulation does not occur. The eSham system was used to mimic sensations of real rTMS. This system produces mild tingling on the scalp underneath the sham rTMS coil, making it difficult in differentiating between real and sham. The amount of electrical stimulation necessary to match real rTMS pulses was determined using an algorithm (parameter estimation by sequential testing). All subjects underwent the sham titration at the beginning of every rTMS session regardless of group assignment. The left prefrontal cortex was the cortical target for rTMS treatment, located using the EEG-10-20 system.
  Other Names: NeoPulse Neotonus Model 3600
  Arms: Both Sham TMS; Sham then Real TMS
Device: Real TMS 4 Hours — Real TMS 4 hours after surgery, first determined resting motor threshold (rMT) by starting with 40% of the machine output and 0.5 Hz stimulus frequency. The coil was positioned over the motor cortex and then adjusted until each pulse results in movement of the right thumb. The machine output was then adjusted to the lowest intensity that reliably produces thumb movement. Parameter estimation by sequential testing was used to determine the amount of machine energy necessary to visibly move the thumb 50% of the time. rMT was assessed before each rTMS treatment. The left prefrontal cortex was the cortical target for rTMS treatment. The EEG-10-20 system was used to locate the prefrontal cortex (F3).
  Other Names: NeoPulse Neotonus Model 3600
  Arms: Both Real TMS; Sham then Real TMS
Device: Sham TMS 4 Hours — Sham TMS 4 hours after surgery used specifically designed rTMS coil that produces auditory signals identical to real (active) TMS coils but is shielded so that actual stimulation does not occur. The eSham system was used to mimic sensations of real rTMS. This system produces mild tingling on the scalp underneath the sham rTMS coil, making it difficult in differentiating between real and sham. The amount of electrical stimulation necessary to match real rTMS pulses was determined using an algorithm (parameter estimation by sequential testing). All subjects underwent the sham titration at the beginning of every rTMS session regardless of group assignment. The left prefrontal cortex was the cortical target for rTMS treatment, located using the EEG-10-20 system.
  Other Names: NeoPulse Neotonus Model 3600
  Arms: Both Sham TMS; Real then Sham TMS

SUMMARY:
The purpose of this research study is to investigate the effects of Transcranial Magnetic Stimulation on pain perception. TMS is a non - invasive technique that uses electromagnetic pulses to temporarily stimulate specific brain areas in awake people (without the need for surgery, anesthetic, or other invasive procedures)

DETAILED DESCRIPTION:
To test whether rTMS over the left prefrontal cortex significantly reduces post-operative pain and PCA use following gastric-bypass surgery relative to sham and an active control, in a mood- independent manner. Note that the active control is still mentioned in the aims and hypotheses, but was apparently removed from the study design.

To determine the effects of timing (one immediately following surgery and one 4 hours later) and dose of TMS (0, 1, or 2 sessions of active rTMS) on post-operative pain and PCA use; To determine the effects of TMS on post-surgical recovery time (time to discharge) and clinical outcomes at 1-month, 3- months and 6-months follow-up. Again an active control is mentioned, though this was removed from the design. It appears that this aspect of the proposal was not edited to reflect the new study design.

In the new design, 108 participants received two 20 minute sessions of 10 Hz rTMS (110% of motor threshold) over the left dorsolateral prefrontal cortex (one immediately following surgery and one 4 hours later). Participants were randomly assigned to receive two sessions of real rTMS, two sessions of sham, 1 real then 1 sham, or 1 sham then 1 real rTMS treatments.

ELIGIBILITY:
Inclusion Criteria:

* Adult gastric by-pass patients 18 to 60 years old

Exclusion Criteria:

* Non gastric by -pass patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2005-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Borckardt, Principal Investigator — Medical University of South Carolina
Locations (1):
- Institute of Psychiatry Brain Stimulation lab, Charleston, South Carolina, United States

REFERENCES:
- [Result] Borckardt JJ, Reeves ST, Kotlowski P, Abernathy JH, Field LC, Dong L, Frohman H, Moore H, Ryan K, Madan A, George MS. Fast left prefrontal rTMS reduces post-gastric bypass surgery pain: findings from a large-scale, double-blind, sham-controlled clinical trial. Brain Stimul. 2014 Jan-Feb;7(1):42-8. doi: 10.1016/j.brs.2013.07.007. PMID 24527503
- See also: Link to Published Manuscript for NCT01861574 (HR 15330) — https://www.ncbi.nlm.nih.gov/pubmed/24527503

RESULTS

PARTICIPANT FLOW:
Groups:
- Both Real TMS: Gastric-Bypass Patients receive Real TMS 45 minutes after gastric-bypass surgery Gastric-Bypass Patients receive Real TMS 4 hours after gastric-bypass surgery
- Sham Then Real TMS: Gastric-Bypass Patients receive Sham TMS 45 minutes after gastric-bypass surgery Gastric-Bypass Patients receive Real TMS 4 hours after gastric-bypass surgery
- Real Then Sham TMS: Gastric-Bypass Patients receive Real TMS 45 minutes after gastric-bypass surgery Gastric-Bypass Patients receive Sham TMS 4 hours after gastric-bypass surgery
- Both Sham TMS: Gastric-Bypass Patients receive Sham TMS 45 minutes after gastric-bypass surgery Gastric-Bypass Patients receive Sham TMS 4 hours after gastric-bypass surgery
Period: Overall Study
Arm/Group | Both Real TMS | Sham Then Real TMS | Real Then Sham TMS | Both Sham TMS
Started | 28 | 25 | 27 | 28
Completed | 28 | 25 | 27 | 28
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Both Real TMS | Sham Then Real TMS | Real Then Sham TMS | Both Sham TMS | Total
Number analyzed (Participants) | 28 | 25 | 27 | 28 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 25 | 27 | 28 | 108
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.21 (11.90) | 45.44 (10.07) | 44.33 (8.96) | 49.89 (12.35) | 47.04 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 19 | 18 | 79
  Male | 7 | 4 | 8 | 10 | 29
Region of Enrollment [Number; unit: participants]
  United States | 28 | 25 | 27 | 28 | 108

OUTCOME MEASURES:

1. Primary Outcome: Patient Controlled Analgesia (PCA) Hydromorphone Usage
Description: PCA pump usage values were reported by concentration in mg/mL. Post operative PCA pump usage was tracked 0-48 hours after surgery. The PCA pump usage was downloaded from the PCA pump after discharge from the hospital and values were reported in mg/mL (concentration in mg/mL). The PCA pump data were averaged over Post-operative hours 0-48 (total PCA pump usage post-operatively) and the mean PCA pump usage was calculated and reported in mg/mL for all groups (4).
Time Frame: Post-Op Hour 0 through 48
Measure: Mean (Standard Deviation); unit: mg/ml
Arm/Group | Both Real TMS | Sham Then Real TMS | Real Then Sham TMS | Both Sham TMS
Number analyzed (Participants) | 28 | 25 | 27 | 28
mg/ml | 11.77 (7.67) | 13.42 (6.92) | 12.66 (7.65) | 9.83 (5.59)

2. Primary Outcome: Sensory Dimension of McGill Pain Questionnaire
Description: Participants completed the McGill Pain Questionnaire-short form (MPQ) at Check Up 1, Check Up 2, Check Up 3, and Check Up 4. Check Up 1 & 2 occurred on Post-Op Day 1. Check Up 1 occurred immediately after surgery. Check Up 2 occurred 4 hours after Check Up 1. Check Up 3 & 4 occurred on Post-Op Day 2, 4 hours apart.
  The MPQ has two pain dimensions: 1.Sensory subscale with 11 words, and 2.Affective subscale with 4 words from the original MPQ. The range of scores for the affective dimension of pain is 0-12.
  The range of scores for the sensory dimension of pain is 0-33. The maximum total score for the sensory dimension is 33.
  Higher scores are indicative of worse pain on the sensory dimension of pain.
Time Frame: Check Up 1, Check Up 2, Check Up 3, and Check Up 4
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Both Real TMS | Sham Then Real TMS | Real Then Sham TMS | Both Sham TMS
Number analyzed (Participants) | 28 | 25 | 27 | 25
units on a scale
  Check up 1 | 6.33 (1.35) | 5.36 (1.06) | 4.8 (0.84) | 5.71 (1.32)
  Check up 2 | 4.5 (0.68) | 5.4 (.94) | 5.03 (0.88) | 5.5 (0.94)
  Check up 3 | 4.72 (0.77) | 5.82 (1.3) | 5.96 (1.19) | 7.07 (1.3)
  Check up 4 | 4.71 (0.88) | 5.62 (0.95) | 8 (1.39) | 8.68 (1.6)

3. Secondary Outcome: Correctly Guessed Assignment Condition at 4 Hours
Description: Participants were asked to guess whether they received real or sham TMS after each rTMS session. The results below report the percentage or participants that correctly guessed TMS Condition after the second TMS treatment, 4 hours after surgery.
Time Frame: After second TMS treatment (Check up 4)
Measure: Number; unit: percentage of participants
Groups:
- All Participants: All 108 participants
Arm/Group | All Participants
Number analyzed (Participants) | 108
percentage of participants | 53

4. Secondary Outcome: Confidence Ratings of Guessing TMS Condition Assignment
Description: After participants guessed their TMS condition; whether they received real or sham TMS, They were then asked to rate the confidence in their guess. Ratings were on a scale of 0-10 where 0=complete guess and 10=absolutely sure.
  Results below include the mean confidence ratings of those that guessed the TMS condition correctly and those that guessed incorrectly.
Time Frame: After Second TMS Treatment (Check up 4)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Correct Guess: 57 of 108 Participants guessed the correct TMS condition
- Incorrect Guess: 51 of 108 Participants incorrectly guessed their TMS condition
Arm/Group | Correct Guess | Incorrect Guess
Number analyzed (Participants) | 57 | 51
units on a scale | 5.40 (3.16) | 6.52 (2.51)

5. Primary Outcome: Affective Dimension of McGill Pain Questionnaire
Description: Participants completed the McGill Pain Questionnaire-short form (MPQ) at Check Up 1, Check Up 2, Check Up 3, and Check Up 4. Check Up 1 & 2 occurred on Post-Op Day 1. Check Up 1 occurred immediately after surgery. Check Up 2 occurred 4 hours after Check Up 1. Check Up 3 & 4 occurred on Post-Op Day 2, 4 hours apart.
  The MPQ has two pain dimensions: 1.Sensory subscale with 11 words, and 2.Affective subscale with 4 words from the original MPQ. The range of scores for the affective dimension of pain is 0-12.
  The maximum total score for the Affective dimension is 12. Higher scores are indicative of worse pain on the affective dimension of pain.
Time Frame: Check Up 1, Check Up 2, Check Up 3, and Check Up 4
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Both Real TMS | Sham Then Real TMS | Real Then Sham TMS | Both Sham TMS
Number analyzed (Participants) | 28 | 25 | 27 | 28
units on a scale
  Check up 1 | 2.33 (0.64) | 0.95 (028) | 1.29 (0.36) | 1.6 (0.4)
  Check up 2 | 1.35 (0.3) | 1.35 (0.4) | 1.64 (0.57) | 1.88 (0.35)
  Check up 3 | 1.08 (0.28) | 1.4 (0.6) | 1 (0.21) | 2.5 (0.53)
  Check up 4 | 0.88 (0.2) | 1.62 (0.43) | 1.86 (0.44) | 3 (0.76)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Both Real TMS | Sham Then Real TMS | Real Then Sham TMS | Both Sham TMS
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/25 | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/25 | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/25 | 0/27 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No